CLINICAL TRIAL: NCT07285811
Title: Whey Protein Dose-response Effect on Daily Glycaemic Excursions in Very Old Individuals With Type 2 Diabetes
Brief Title: GLycaemic Outcomes With Whey Protein in ageING
Acronym: GLOWING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: RG_24-052
Record Dates: First submitted 2025-11-18; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Whey Proteins

STUDY DESIGN:
Intervention Model Description: Placebo-controlled partial crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pre-meal low dose whey protein (Active Comparator): Low whey protein dose administration before meals
  Interventions: Dietary Supplement: Glycaemic control with whey protein; Dietary Supplement: Glycaemic control with different doses of whey protein
- pre-meal moderate dose whey protein (Active Comparator): Moderate whey protein dose administration before meals
  Interventions: Dietary Supplement: Glycaemic control with whey protein; Dietary Supplement: Glycaemic control with different doses of whey protein
- pre-meal protein-free placebo (Placebo Comparator): protein-free placebo administration before meals
  Interventions: Dietary Supplement: Glycaemic control with whey protein

INTERVENTIONS:
Dietary Supplement: Glycaemic control with whey protein — Comparing pre-meal supplementation of whey protein to protein-free placebo.
Dietary Supplement: Glycaemic control with different doses of whey protein — Comparing pre-meal supplementation of moderate whey protein to a low dose of whey protein.
  Arms: pre-meal low dose whey protein; pre-meal moderate dose whey protein

SUMMARY:
The goal of this placebo-controlled, partial crossover design study is to identify the impact of consuming whey protein before meals on free-living glucose control in older adults living with type 2 diabetes.

The primary specific objective is to determine the effect of a thrice daily whey protein pre-meal supplementation at two doses, on glucose excursions over a 7-day free-living period in adults aged 75-90 years of age, living with type 2 diabetes, compared with a non-protein placebo.

Participants will consume the whey protein and placebo for 7 days each, before each meal. All participants will consume the placebo and one of two doses of whey protein, in a randomised order.

DETAILED DESCRIPTION:
Within the study, the researchers will look at the effect of supplemental whey protein at moderate and low doses in comparison to each other and a protein-free placebo on glycaemic control in older adults aged between 75-90 years of age, living with type 2 diabetes.

Glycaemic control (glucose excursions) will be monitored under free-living conditions over a 7-day period using continuous glucose monitors (CGMs). Participants will be randomised to consume one of the two whey protein doses as well as the protein-free placebo on a separate 7-day period. The order of consuming whey protein or the protein-free placebo will be randomised and counterbalanced. This study is under the evidence that in younger people living with type 2 diabetes, a moderate dose of whey protein improves glucose time in range and lessens extreme postprandial glucose excursions.

Participants will be free to consume their typical diet over this period, where the researchers will provide a diet diary for participants to enter in all foods and drinks they consume over this time period, as well as document the ingestion of the supplement before each main meal.

During an acute feeding period on the first ingestion of each supplement (start of each 7-day phase), the researchers will evaluate rates of gastric emptying, glucose and insulin concentrations and hormonal appetite markers through blood draws, as well as perceived appetite responses through visual analogue scales. This will be in a research kitchen where participants will consume the supplement and a controlled mixed meal afterwards to monitor excursions in appetite response and glycemia. The researchers will also investigate the impact of pre-meal protein feeding on renal markers following each 7-day phase via urine collection.

ELIGIBILITY:
* Male or female
* 75-90 years old
* Type 2 Diabetes (confirmed with glycated haemoglobin (HbA1c) >6.5% in clinic or in SportExR)
* Stable body mass (body mass index (BMI) ≤40kg/m2)
* Generally healthy, assessed via a General Health Questionnaire (GHQ)
* Some residual beta-cell activity (confirmed with urine test on induction)
* Normal or moderately increased albuminuria (needs to be below 300mg/g)
* Normal, mildly or moderately decreased glomerular filtration rate (GFR) (needs to be above 45ml/min/1.732).
* Able and willing to attend SportExR a total of 5 times: 1 induction and 2 testing visits and 2 return check-up visits.

Exclusion Criteria:

* <75 years old and over 90 years of age
* Currently on fast-acting insulin therapy (i.e., Humalog)
* Confirmed uncontrolled diabetes (HbA1C >10% or 85mmol/mol).
* Currently on GLP-1 therapy
* Habitual smoker or vaper
* Veganism
* Lactose or dairy intolerance
* Coeliac or gluten intolerance
* History of gastrointestinal disease
* Experienced a hyperglycaemic or hypoglycaemic event requiring treatment in the past 12 months
* Recent Ischemic stroke (<3 months).
* Use of anticoagulants (e.g. warfarin, rivaroxaban)
* Considered unwilling or unable to comply with the study protocol requirements by the research team

Ages: 75 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of changes in free-living glycaemic control | 7 days, two occasions
  Time spent in normal glucose range, under free-living conditions with pre-meal supplementation (measured by continuous glucose monitors)
Changes in postprandial glucose concentrations in blood | 4 hours, two occasions
  Amplitude of post-meal blood glucose following supplement(s) and controlled meal
Concentrations of insulin postprandially in blood | 4 hours, two occasions
  Insulin appearance in blood following supplement(s) and controlled meal

SECONDARY OUTCOMES:
Concentrations of amino acids postprandially in blood | 4 hours, two occasions
  Total amino acid appearance in blood following supplement(s) and controlled meal
Concentrations of postprandial appetite hormones | 4 hours, two occasions
  Postprandial appetite hormone concentrations in blood following supplement(s) and controlled meal
Rate of gastric emptying | 4 hours, two occasions
  Rate of gastric emptying using acetaminophen appearance in the blood following its consumption with supplement(s) and controlled meal.
Changes in renal function markers after each 7-day phase | 2 urine samples, 2 occasions
  Measurement of markers of renal function from urine following each 7-day phase
Assessment of nitrogen balance from urine after each 7-day phase | 24 hours, two occasions
  Nitrogen balance from 24-hour urine collection after each 7-day phase
Measurement of blood lipid concentration | 1 blood draw (obtained from the first blood draw as part of 4 hour visit)
  Total cholesterol measurement in blood at rest
Optional qualitative assessment of perceptions to supplementation | 60 minutes
  Optional interview for participants to share perceptions of pre-meal supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Breen, PhD, Principal Investigator — University of Birmingham and University of Leciester
Locations (2):
- United Kingdom (2):
  - School of Sport, Exercise and Rehabilitation Sciences, University of Birmingham, Birmingham, West Midlands
  - Heartlands Hospital, Birmingham